CLINICAL TRIAL: NCT06447714
Title: A Prospective Cohort Study on the Correlation Between Patient Cotinine Levels and Intracranial Unruptured Aneurysm Wall Enhancement Based on High-resolution Magnetic Resonance Imaging
Brief Title: A Study on the Correlation Between Cotinine Levels and Aneurysm Wall Enhancement on HRMRI.
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LC2024ZD028
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cotinine Levels; Arterial Aneurysm Wall Enhancement on HRMRI
MeSH Terms: interventions — Smoke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient plasma sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No aneurysm wall enhancement: The aneurysm wall did not show enhanced signal on high-resolution magnetic resonance imaging.
- Aneurysm wall enhancement: The aneurysm wall shows enhanced signal on high-resolution magnetic resonance imaging.
  Interventions: Behavioral: smoke

INTERVENTIONS:
Behavioral: smoke — cotinine detection
  Groups: Aneurysm wall enhancement

SUMMARY:
This study aims to collect clinical, laboratory, and imaging data from patients with unruptured intracranial aneurysms, and collect blood or urine samples for cotinine testing. The enrolled patients underwent high-resolution magnetic resonance angiography to detect whether the intracranial aneurysm wall was enhanced and classify the degree of enhancement. The purpose is to study the correlation between arterial aneurysm wall enhancement and cotinine levels

DETAILED DESCRIPTION:
This study aims to explore the relationship between cotinine levels and the risk of intracranial aneurysm rupture by collecting imaging features and patient cotinine levels of unruptured intracranial aneurysms on high-resolution magnetic resonance imaging, combined with the prognosis of patients with aneurysms. Previous studies have shown that the risk of intracranial aneurysm rupture in patients is related to the enhancement of the aneurysm wall on high-resolution magnetic resonance imaging. Therefore, this study included patients who met the inclusion criteria for high-resolution magnetic resonance imaging and cotinine testing, and followed up on the imaging characteristics, prognostic scores, and aneurysm occlusion rate of arterial aneurysms in patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, male or infertile female;
* Diagnosed as IA (intracranial aneurysm) through CTA, MRA, or DSA; And it is suitable for endovascular intervention treatment
* The patient and/or their legal representative or guardian fully understand the research purpose, voluntarily participate and sign informed consent Books;
* Patients willing to cooperate with high-resolution magnetic resonance imaging.
* Patients willing to follow up and evaluate according to clinical research protocol requirements

Exclusion Criteria:

* AVM (arteriovenous malformation), Moyamoya disease, or DAVF (dural arteriovenous fistula) related aneurysms;
* Patients with contraindications for high-resolution magnetic resonance imaging;
* Participants in clinical trials of other drugs or medical devices;
* Patients with severe underlying diseases and extremely poor clinical conditions who cannot tolerate general anesthesia surgery;
* Patients with poor compliance and inability to cooperate with follow-up;
* Possible or clear history of severe allergy to contrast agents;
* Patients with a life expectancy of less than 2 years;
* Women who are breastfeeding and preparing for pregnancy during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed intracranial unruptured aneurysm patient through DSA/MRA/CTA examination
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
High resolution MRI aneurysm features | 1 year
  Enhancement grade was defined as follows: grade 0 for none enhancement, grade 1 for focal enhancement, involved the neck, the intermediate portion, the dome, or a bleb;grade 2 for thin annular enhancement (maximum thickness≤1 mm) , grade 3 for thick annular enhancement(maximum thickness>1 mm) .
postoperative 12 month mRS score | 1 year
  MRS score definition: The MRS score, also known as the Modified Rankin Scale, is a scale used to evaluate the neurological recovery status of stroke patients. It is divided into seven levels, Level 0: completely asymptomatic. Level 1: Despite symptoms, without obvious disabilities, able to complete all frequently engaged work and activities.
  Level 2: Mild disability, unable to complete all work and activities, but able to handle personal affairs without the need for assistance from others.
  Level 3: Moderate disability, requiring assistance from others to walking without assistance.
  Level 4: Severe disability, unable to walk without the help of others, unable to take care of one's own needs.
  Level 5: Severe disability, bedridden, urinary and fecal incontinence, requiring continuous care, and requiring multiple 24-hour care from others.
  Level 6: Death. The higher the mRS score, the worse the patient's prognosis.
postoperative 12 month aneurysm occlusion rate | 1 year
  Raymond classification, grade I: complete embolism; Grade II: residual aneurysm neck; Grade III: Residual aneurysm cavity. The higher the Raymond grade, the lower the successful embolization rate of the patient's aneurysm.
  OKM classification is A1/A2/A3; B1/B2/B3; C1/C2/C3; D/Unsuccessful (note: A, B, C, D represent the volume of contrast agent filled aneurysm, A represents>95%, B represents 5-95%, C represents<5%, D represents no filling). 1, 2, and 3 represent the degree of contrast agent retention in the aneurysm, 1 represents only retention in the arterial phase, 2 represents retention continuing into the capillary phase, and 3 represents still retention in the venous phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China